CLINICAL TRIAL: NCT03599635
Title: Ultrasound-guided Pec Infiltration With Liposomal Bupivacaine for Breast Surgery: A Prospective Randomized Study
Brief Title: Pec Infiltration With Liposomal Bupivacaine for Breast Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANES-2017-25584
Record Dates: First submitted 2018-06-20; First posted 2018-07-26 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- liposomal bupivacaine (Experimental): These patients will receive liposomal bupivacaine for a pectoralis block infiltration by the anesthesiologist.
  Interventions: Drug: liposomal bupivacaine
- bupivacaine (Active Comparator): These patients will receive incisional bupivacaine infiltration by the surgeon.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: liposomal bupivacaine — Experimental
  Arms: liposomal bupivacaine
Drug: Bupivacaine — Active Comparator
  Arms: bupivacaine

SUMMARY:
The purpose of this study is to compare pain control after breast surgery using either liposomal bupivacaine or bupivacaine when infiltrated during an ultrasound guided pectoralis 1 and 2 block. Both medications, liposomal bupivacaine and bupivacaine, are standard of care in these types of surgeries.

DETAILED DESCRIPTION:
For the Pec infiltration, the patient will be in the supine position. The pectoralis major and pectoralis minor muscle layers will be identified via ultrasound. Using sterile technique, a nerve block needle will be inserted and advanced under ultrasound guidance until it is below the fascial covering of the pec minor muscle layer. Gentle aspiration for air or blood will be performed in 5cc incremental doses. Then injection of 10 mL of bupivacaine 0.25% with epinephrine 1:200,000 and 10mL of a mixture of liposomal bupivacaine and saline (5 mL liposomal bupivacaine and 5 mL saline) for a total injection for pec 1 block of 20 mL. For each 5cc of local anesthetic injected, aspiration will be performed. Upon completion of the injection the needle will be removed. The investigators will then use the ultrasound probe to identify the second rib on anterolateral chest wall and move the probe to the 4th rib. Here the investigators will identify the pec minor and serratus anterior muscles. They will advance their needle under ultrasound-guidance beneath pec minor and above serratus anterior. Here an injection 10 mL 0.25% bupivacaine with epinephrine 1:200,000 followed by 20 mL mixture of 15 mL liposomal bupivacaine and 5 mL saline for a total volume of 30ml for Pec 2. block will occur.

Upon completion of the injection, the needle will then be removed and the patient will be monitored in the preoperative area until he/she is brought into the operating room for their procedure.

If deemed necessary for coverage the surgeon will be allowed to inject additional local anesthetic up to a maximum of 40 mL of 0.25% bupivacaine. This will be noted in the chart.

For the surgeon infiltration, the patient will be brought directly to the operating room where intraoperative anesthetic with an opioid-sparing MAC technique will be provided as described below. Just prior to the skin incision, 0.25% bupivacaine will be used to infiltrate the dermis and subcutaneous space in the proposed incision. Throughout the procedure, additional incisional bupivacaine infiltration into the surrounding tissues will be performed as needed for local anesthesia. A total of up to 30 mL of 0.25% bupivacaine will be divided equally for the two sides of the incision. An additional 5 mL of 0.25% bupivacaine will be infiltrated into the pectoralis major muscle at the deep margin of resection. Accidental intravascular injection is minimized by continuous needle movement and frequent aspiration.

The following vital signs will be monitored throughout the procedure: Heart rate, blood pressure, oxygen saturation, and respirations, and patient's state of consciousness. The investigators will monitor the patient until they are brought to the operating room for surgery.

All patients will receive multimodal analgesia in the preoperative area. They will receive 975 mg of oral acetaminophen and 300 mg of gabapentin orally prior to surgery. 30 mg of ketorolac will be given just prior to closure in the operating room.

The intraoperative anesthetic will be an opioid-sparing MAC anesthetic. Patients will receive IV midazolam 0-2 mg followed by 40-100mg of IV lidocaine, and followed by a propofol infusion with 2 mg/ml of ketamine. Opioids will be avoided unless HR or BP increases by 20 % above baseline. Then only short acting opioids (fentanyl) will be given. If patients are unable to tolerate procedure under MAC they would be converted to a general anesthetic with an laryngeal mask airway (LMA).

In the recovery room if the patient experiences pain greater than 5/10 they will receive either IV or oral pain medications. If pain score is less than 5 patients will get non opioid medications unless the patient desires an opioid medication.

When the operation is complete the patient will either be brought to the PACU or Phase II. Each day a member of the research team will call and evaluate the patient for signs of complications and ask the patient their minimum and maximum pain score (scores will be evaluated at 1 hr, 2 hr, 6hrs, 24hrs, 48hrs, 72hrs). They will record daily opioid use, any modality related complications, how many phone calls were made regarding pain control and modality related complications. At time period 72 hours a Quality of recovery survey (see appendix) and OBAS (see appendix) survey will be presented to patient.

At 3 months, 6 months, and 12 months patients will be called to answer a survey with regards to chronic pain.

Patients will be instructed to take acetaminophen 1000 mg every 8 hours while at home and alternate that every four hours with ibuprofen 800 mg every 8 hours. They will be given a prescription of opioid pain medications either oxycodone or hydrocodone and will be instructed to take as needed for pain.

ELIGIBILITY:
Inclusion Criteria:

* • All patients undergoing partial mastectomy procedures.

  * Ages 18-75

Exclusion Criteria:

* • Patient on chronic anticoagulation

  * Pregnant women
  * Non-english speaking patients
  * Any individuals who are unable to give informed consent
  * Any individual with diminished capacity to give informed consent
  * Allergy to local anesthetics
  * Patients who remain intubated overnight after surgery or who are unable to provide information regarding their pain immediately postoperatively
  * Daily use of opioid for more than three weeks
  * Significant liver disease, defined as liver enzymes greater than 3x the upper limit of normal
  * Lack of patient cooperation including those patients who refuse a MAC anesthetic
  * Contraindication to regional anesthesia

    * Infection at injection site
    * Inability to guarantee sterile equipment or sterile conditions for the block
    * Patient refusal
    * Severe Coagulopathy or bleeding disorder

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Habeck, MD, Principal Investigator — University of Minnesota
Locations (1):
- M Health Ambulatory Surgery Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EVEN Number = PEC Block: Midazolam 0-2 mg IV. NO Fentanyl. 20mL injection below pec minor fascia 10mL 0.25% bupivacaine with epinephrine 1:200,000 followed by 10mL of a mixture of 5mL liposomal bupivacaine and 5mL saline.
- ODD Number = Surgeon Infiltration: 30mL injection beneath pec minor and above serratus anterior or if unable to visualize the serratus/pec minor border will inject under the serratus anterior at the 4th rib 10 mL 0.25% bupivacaine with epinephrine 1:200,000 followed by 20 mL mixture of 15 mL liposomal bupivacaine and 5 mL saline.
Period: Overall Study
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Started | 56 | 55
Completed | 56 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 45 | 86
  >=65 years | 15 | 10 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 2 | 7
  White | 43 | 44 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Use
Description: Description: To determine if liposomal bupivacaine Pec infiltration provides decreased peri-operative opioid usage when compared to incisional bupivacaine infiltration.
Time Frame: time from end of surgery through 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
mg | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

2. Secondary Outcome: Maximal Pain Scores - 1 Hour
Description: total additive maximal patient pain scores measured using a numerical rating scale pain score 0-10 at time points 1 hour, 2, hours, 6 hours, 24 hours, 48 hours, and 72 hours. Higher pain score is worse pain score.
Time Frame: 1 hour
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 1.0 [0.0 to 4.0] | 2.0 [0.0 to 4.0]

3. Secondary Outcome: Maximal Pain Scores - 2 Hours
Description: as for outcome 2
Time Frame: 2 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 1.5 [0.0 to 3.0] | 1.0 [0.0 to 3.0]

4. Secondary Outcome: Maximal Pain Scores - 6 Hours
Description: as for outcome 2
Time Frame: 6 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 1.0 [0.0 to 2.3] | 2.0 [1.0 to 3.5]

5. Secondary Outcome: Maximal Pain Scores - 24 Hours
Description: as for outcome 2
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 1.0 [0.0 to 3.0] | 2.0 [1.0 to 4.0]

6. Secondary Outcome: Maximal Pain Scores - 48 Hours
Description: as for outcome 2
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 1.0 [0.0 to 3.0] | 2.0 [1.0 to 3.0]

7. Secondary Outcome: Maximal Pain Scores - 72 Hours
Description: as for outcome 2
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 1.0 [0.0 to 2.0] | 1.0 [0.0 to 3.0]

8. Secondary Outcome: Improved Quality of Recovery Score
Description: To determine if a pectoralis 1 and 2 block with liposomal bupivacaine improves quality of recovery score post-operatively when compared to incisional bupivacaine infiltration. The scale used was QR15 with 0 to 150 scale; 0 is non of the time/poor, 150 all of the time/excellent.
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 142.0 [132.0 to 148.0] | 138.0 [130.0 to 143.5]

9. Secondary Outcome: Effect in Patients With Breast Surgery
Description: To observe the effect on chronic postoperative pain in patients who have breast surgery, measured with the Overall Benefit of Analgesia Score (OBAS), where 0 is minimal pain and 4 is maximum pain.
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
Number analyzed (Participants) | 56 | 52
score on a scale | 2.0 [0.0 to 4.0] | 4.0 [1.0 to 5.0]

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | EVEN Number = PEC Block | ODD Number = Surgeon Infiltration
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55
Other Adverse Events (participants affected / at risk) | 7/56 | 6/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVEN Number = PEC Block (N=56) | ODD Number = Surgeon Infiltration (N=55)
Nausea/ Vomiting (Gastrointestinal disorders) | 7 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/35/NCT03599635/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT03599635/ICF_001.pdf